CLINICAL TRIAL: NCT06823050
Title: A Prospective, Multicenter, Phase II Clinical Study on the Treatment of Unresectable Advanced Hepatocellular Carcinoma with the DEB-TACE (drug-loaded Microsphere Transcatheter Arterial Chemoembolization) Combined with Hepatic Artery Perfusion of Raltitrexed and Oxaliplatin (SALOX-HAIC) Regimen
Brief Title: A Prospective, Multicenter, Phase II Clinical Study on the Treatment of Unresectable Advanced HCC with DEB-TACE Combined with SALOX-HAIC
Status: Not yet recruiting | Type: Observational
Sponsor: Xuhua Duan (Other)
Responsible Party: Sponsor-Investigator, Xuhua Duan, Associate Professor, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Other Study IDs: 2025-KY-0112-001
Record Dates: First submitted 2025-02-07; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- DEB-TACE+ SALOX-HAIC+Apatinib+Carilizumab: Drug-eluting bead transarterial chemoembolization combined with SALOX-HAIC sequential Apatinib and Carilizumab

SUMMARY:
The aim of this study is to clarify the safety and efficacy of DEB-TACE combined with SALOX-HAIC in the treatment of unresectable advanced primary liver cancer. To determine whether this therapy can prolong the indicators such as PFS, TTP, OS, ORR, and DOR.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient with unresectable HCC who strictly meet the clinical diagnostic criteria of the Guidelines for Diagnosis and Treatment of Primary Liver Cancer (2024 Edition) or who have been confirmed by histopathology or cytology, There was at least one measurable lesion (according to the requirements of mRECIST 1.1, the spiral CT scan diameter of the measurable lesion was ≥10mm or the short diameter of enlarged lymph node was ≥15mm).

  2. CNLC Ib-IIIa；BCLC：A-C 3. Patient age between 18 and 80，male or female. 4. ECOG 0-1. 5.Expected life span ≥ 3 months. 6. No history of severe comorbidities, such as hypertension, coronary heart disease, and mental illness, and no history of severe allergies.

  7. Child-Pugh A-B. 8.The laboratory tests meet the following requirements: platelets ≥ 50×109/L; hemoglobin ≥ 9g/dL; white blood cells ≥ 4×109/L; neutrophils ≥ 1.5×109/L; serum total bilirubin ≤ 1.5 times the upper limit of normal value (ULN), transaminases (ALT, AST) ≤ 5 times ULN; creatinine ≤ 1.5 times ULN; urine routine test shows that urine protein < 2+; for patients whose urine routine test at baseline showed urine protein ≥ 2+, 24-hour urine collection should be conducted and the 24-hour urine protein quantification should be < 1g; international normalized ratio (INR) or activated partial thromboplastin time (APTT) ≤ 1.5 times ULN.

  9. HBV DNA<2000 IU/ml. 10. Women of childbearing age must undergo a pregnancy test within 7 days prior to enrollment.

  11. Patients sign informed consent, good compliance, cooperate with treatment.

Exclusion Criteria:

* 1. Imaging examinations were conducted for HCC patients with large liver tumors (≥60% of liver volume), or carcinoma thrombus in main portal vein (occupying ≥50% of vascular diameter), or carcinoma thrombus invading mesenteric vein or inferior vena cava, or significant arteriovenous/venous fistula.

  2. Before participating in this study, she had received local treatment such as TACE, external radiotherapy and radioactive particle implantation, and had undergone systemic chemotherapy, oral liver cancer targeting drugs (Sorafenib, Lenfacitinib, Apatinib) and immunotherapy such as PD-1/PD-L1/CDLA-4.

  3. Diffuse liver cancer patients. 4. Patients with grade Ⅱ or above myocardial ischemia or myocardial infarction, poorly controlled arrhythmias (including QTc interval ≥450ms for men and 470ms for women.

  5. A history of gastrointestinal bleeding within the past 6 months or a definite tendency to gastrointestinal bleeding.

  6. Abnormal clotting function, bleeding tendency or receiving thrombolytic or anticoagulant therapy.

  7. Patients with central nervous system metastases or known brain metastases. Co-infected patients with HIV; Pregnant or lactating patients. Patients preparing for liver transplantation (other than those with previous liver transplantation.

  8. Systemic failure, estimated survival time <3 months. 9. Severe renal dysfunction. 10. The patients could not complete the treatment plan due to various reasons, and lost control within three months after enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: unresectable advanced HCC
Sampling Method: Non-Probability Sample
Enrollment: 59 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Time from the first DEB-TACE treatment to either radiological progression or death or up to 24 months

SECONDARY OUTCOMES:
Overall survival (OS) | Time Frame: Time from the first DEB-TACE treatment to death or up to 24 months
Objective response rate (ORR) | 1, 3, 6,12,18,24 months after the first DEB-TACE treatment, up to death or 24 months, whichever came first.
Disease control rate (DCR) | 1, 3, 6,12,18,24 months after the first DEB-TACE treatment, up to death or 24 months, whichever came first
Time to Progression (TTP) | Time from the first DEB-BACE treatment to either radiological progression up to 24 months

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Deng zhou People's Hospital, Dengzhou, Henan
  - The Second People's Hospital of Jiaozuo, Jiaozuo, Henan
  - Huai He Hospital of Henan University, Kaifeng, Henan
  - Luo Yang Central Hospital, Luoyang, Henan
  - First People's Hospital of Shangqiu, Shangqiu, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Zhou Kou Central Hospital, Zhoukou, Henan